CLINICAL TRIAL: NCT01377142
Title: Vaginal Uphold Hysteropexy and Laparoscopic Sacral Hysteropexy for the Treatment of Uterovaginal Pelvic Organ Prolapse
Acronym: VAULT
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: The Christ Hospital (Other); Medstar Health Research Institute (Other); Providence Healthcare (Other); Stanford University (Other); Women and Infants Hospital of Rhode Island (Other); Greater Baltimore Medical Center (Other); University of North Carolina (Other)
Responsible Party: Sponsor
Other Study IDs: 11-409
Record Dates: First submitted 2011-06-10; First posted 2011-06-21 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Pelvic Organ Prolapse
Keywords: Uterovaginal prolapse; hysteropexy; mesh
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Laparoscopic sacral hysteropexy: Laparoscopic sacral hysteropexy is performed laparoscopically with or without robotic assistance
  Interventions: Device: Laparoscopic sacral hysteropexy
- Vaginal mesh hysteropexy: Vaginal Mesh Hysteropexy using the Uphold device which includes Sacrospinous Ligament Fixation
  Interventions: Device: Vaginal mesh hysteropexy

INTERVENTIONS:
Device: Laparoscopic sacral hysteropexy — Laparoscopic sacral hysteropexy is performed laparoscopically with or without robotic assistance
  Groups: Laparoscopic sacral hysteropexy
Device: Vaginal mesh hysteropexy — Uphold device used which includes sacrospinous ligament fixation
  Groups: Vaginal mesh hysteropexy

SUMMARY:
The purpose of this study is to evaluate surgical success or failure one year after surgery for pelvic organ prolapse.

DETAILED DESCRIPTION:
This will be a prospective parallel cohort study comparing a laparoscopic sacral hysteropexy (LSHP) to a vaginal Uphold hysteropexy (VUHP). Symptomatic and anatomic improvement of pelvic organ prolapse will be evaluated at 3 months and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Desires surgical treatment for uterovaginal prolapse.
* Symptomatic stage II-IV POP including:
* cystocele (AA or BA > or = 0) by POP-Q and
* apical descent below the mid-vagina (point C > -(TVL / 2)) by the POP-Q and
* a positive response to questions 3 of the PFDI 20: Do you usually have a bulge or something falling out that you can see or feel in the vaginal area? (Appendix A)
* Eligible for and undergoing one of the following procedures: laparoscopic sacral hysteropexy (LSHP) or Vaginal Uphold hysteropexy (VUHP)
* Female age 40 to 75.
* Completed childbearing confirmed by subject or practicing reliable form of birth control defined as permanent sterilization, hormonal contraception, abstinence, IUD.
* Normal size uterus (length less than 10 cm) on bimanual exam or ultrasound within the past 6 months.

Exclusion Criteria:

* Prior hysterectomy.
* Patient with synthetic material placed to augment previous pelvic organ prolapse repair. (previous prolapse repair without synthetic mesh is acceptable).
* Current vaginal or pelvic foreign body complications (including but not limited to erosion, fistula, abscess). This includes foreign bodies of any type (e.g. synthetic and biologic including allograft, xenograft).
* Desires hysterectomy at the time of prolapse repair.
* Cervical elongation with anticipated need for cervical shortening at the time of prolapse repair as determined by surgeon.
* History of cervical dysplasia (diagnosed within the past 5 years) or increased risk of cervical dysplasia (HIV, immunocompromise, DES exposure), chronic pelvic pain, uterine abnormalities (symptomatic uterine fibroids, polyps, endometrial hyperplasia, cancer) or any uterine disease that would preclude prolapse repair with uterine preservation in the opinion of the surgeon.
* Any postmenopausal bleeding in the past 12 months (regardless of endometrial biopsy or ultrasound results) or any postmenopausal bleeding more than 12 months prior without adequate evaluation in the opinion of the investigator.
* Premenopausal women with menstrual issues including irregular bleeding, menorrhagia, dysmenorrhea,
* Pregnancy (confirmed before surgery with a pregnancy test).

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult women with symptomatic uterovaginal prolapse planning to undergo laparsocopic sacral hysteropexy or vaginal uphold hysteropexy
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2011-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be surgical "success" or "failure" as a dichotomous outcome 1 year after surgery. Subjects will be considered a success if they meet the definitions of anatomic cure and deny vaginal bulging symptoms. | 12 months
  Anatomic sure is defined as cervix above mid-vagina, and no prolapse beyond the hymen and no surgical treatment for pelvic organ prolapse or pessary use.
  Symptomatic cure is defined as the absence of vaginal bulge symptoms as indicated by a negative response question 3 of the pelvic floor distress inventory- 20.

SECONDARY OUTCOMES:
Anatomic outcomes | 12 months
  Evaluation of the anterior and posterior walls using point Aa, Ba, Ap and Bp, C, posterior fornix D and total vaginal length TVL; evaluate the size of the genital hiatus and perineal body; evaluation of cervical elongation and record any additional surgical procedures for anterior and posterior vaginal wall prolapse.
Symptomatic improvement | 3months and 12 months
  Relief of symptoms of pelvic floor disorders, including incontinence, voiding dysfunction, pelvic organ prolapse, fecal incontinence defecation disorders and sexual dysfunction using validated instruments collected postoperatively at 3 months, and 1 year.
Shortterm morbidity | 6 weeks, 3 months, 12 months
  We will compare the treatment groups with respect to perioperative morbidity and mortality. Perioperative morbidity will be recorded at completion of surgery and at hospital discharge. Postoperative morbidity will be recorded at any time after discharge- 6 weeks, 3 months and 1 year and all adverse events will be documented. Perioperative measures of morbidity will include operative time, estimated blood loss, and complications. Length of hospital stay will also be recorded. Complications will be categorized using the Dindo surgical complication grading scale.
Pain and functional activity | 6 weeks and 6 months
  Postoperative pain- subjects will complete the modified surgical pain scale and a diary of pain medication use preoperatively, then daily for two weeks after surgery, then again at 6 weeks postoperatively. Postoperative functional activity level- subjects will complete the activity assessment scale which measures postoperative functional activity preoperatively, 2 weeks, 6 weeks and 6 months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Robert E Gutman, MD, Principal Investigator — Medstar Health Research Institute
Locations (8):
- United States (7):
  - Stanford University, Stanford, California
  - Washington Hospital, Washington D.C., District of Columbia
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - UNC, Chapel Hill, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Women & Infant's Hospital, Providence, Rhode Island
- Providence Healthcare, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No